CLINICAL TRIAL: NCT06915259
Title: Doula Model of Care, A Randomized Controlled Trial
Brief Title: Doula Model of Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Principal Investigator, Sindhu Srinivas, MD, Executive Director, Hospital of the University of Pennsylvania Cedar Avenue, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 857762
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Perinatal; Morbidity; Mental Health
Keywords: Doula; community models of care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants will continue to receive prenatal, labor and delivery, and postpartum care as they normally would if not in the study. Patients who seek doula services on their own will be allowed to do so
- Doula Model of Care (Experimental): Participants will be offered to receive services by the certified doula. The doula will provide emotional support, prenatal support, intrapartum support and will facilitate the receipt of postpartum health care for the patient.
  Interventions: Other: Doula Model of Care

INTERVENTIONS:
Other: Doula Model of Care — Doula model of care is defined as emotional support, prenatal support, intrapartum support, and postpartum support provided to the birthing individual by a certified doula.
  Arms: Doula Model of Care

SUMMARY:
The goal of this randomized controlled intervention trial is to determine if an integrated partnership between a birth worker/community support organization and the Hospital of the University of Pennsylvania (HUP), will improve both the experience and outcomes for Black birthing people.

The main question it aims to answer is whether an integrated partnership between a birth worker/community support organization and the Hospital of the University of Pennsylvania (HUP) will mitigate bias and mistrust thereby improving both the experience and outcomes for Black birthing people, assessed by the primary outcome of depression score.

Participants will be randomized to Doula care (receive 2 prenatal visits, continuous intrapartum support, and 2 postpartum visits with a certified doula) or standard of care (receive prenatal care, labor and delivery, and postpartum care as they normally would if not in the study) and followed through 6 weeks postpartum.

DETAILED DESCRIPTION:
Integrated bi-directional partnerships between birthing facilities, health care providers and community leaders and community birth support persons, such as doulas, is critical to improving health equity and maternal outcomes. This study is partnering with a birth worker/community support organization, with a mission to celebrate Black motherhood and influence favorable outcomes in Black Maternal Health by promoting a community-empowered model of care.

The United States has one of the largest racial and ethnic disparities in pregnancy-related morbidity and mortality of industrialized nations. Black, Indigenous and other people of color (BIPOC) patients have a 2-3 times higher risk of pregnancy-related mortality compared to white patients. For every maternal death, over 100 patients experience a severe maternal morbidity, which is a life-threatening complication during their delivery hospitalization, resulting in over 50,000 women and birthing people experiencing one of these events every year in the U.S. (with the majority occurring in BIPOC patients). These disparities are even more pronounced in the city of Philadelphia, the poorest of the nation's top ten largest cities. A recent report from the Philadelphia Maternal Mortality Review Committee identified 80% of mortalities were among BIPOC patients and 80% of those mortalities had identified social and structural barriers, including, but not limited to, mental health issues, substance use disorders and lack of prenatal care. Integrated bi-directional partnerships between birthing facilities, health care providers and community leaders and community birth support persons, such as doulas, is critical to improving health equity and maternal outcomes. While doulas and other community organizations partner with some birthing providers, the way in which this occurs is variable and the most effective model for integration through the pregnancy continuum has not been determined. Results from previous studies show the importance of implementing community models of care throughout the pregnancy continuum that will mitigate bias, mistrust, and mistreatment thereby improving both the experience and outcomes specifically and especially for Black birthing people.

The study will test the hypothesis that an integrated partnership between a birth worker/community support organization and the Hospital of the University of Pennsylvania (HUP) will mitigate bias and mistrust thereby improving both the experience and outcomes for Black birthing people at HUP. Within this study, the investigators will determine the effectiveness of this integrated partnership in reducing maternal depression score at 6 weeks postpartum. Self-efficacy, perceived trust of care providers, stress, birth satisfaction, and obstetric outcomes will also be assessed. Patients will be randomized (n=230) to Doula care (receive 2 prenatal visits, continuous intrapartum support, and 2 postpartum visits with a certified doula) or standard of care (receive prenatal care, labor and delivery, and postpartum care as they normally would if not in the study) and followed through 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients who self-identify (as seen on Chart) as Black
* Ages 16-55
* Currently pregnant and in second trimester (gestational age between 13-30 weeks)
* Plan to deliver at HUP
* Patients must be able to read and understand English
* Participants must be willing and able to sign the informed consent form

Exclusion Criteria:

* Unable to provide written consent by being unable to read or sign informed consent.
* PI Discretion

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postpartum Depression Scale (EPDS) score | After delivery up to 6 weeks postpartum
  Scores from the validated EPDS screening tool will be calculated using standard scoring criteria for each of the 10 items. A score of 9 or greater or indication of suicide ideation will be used to indicate a positive depression screen

SECONDARY OUTCOMES:
Obstetric outcomes: Mode of delivery | At delivery
  Vaginal or cesarean
Obstetric outcomes: Preterm birth less than 37 weeks | At delivery
  Preterm delivery defined as less than 37 weeks
Obstetric outcomes: Preterm birth less than 34 weeks | At delivery
  Preterm delivery defined as less than 34 weeks.
Self-efficacy | Post-randomization to 6 weeks postpartum
  Self efficacy assessed by the PROMIS General Self-efficacy scale, 10-item scale assessing confidence in ability to deal effectively with a variety of stressful situations. Survey to be completed at randomization and at 6 weeks post partum. The PROMIS General Self-Efficacy measure uses a T-score system, where 50 represents the average for the general population and a standard deviation of 10. A higher T-score indicates greater self-efficacy.
Person centered prenatal care survey for people of color | After delivery up to 6 weeks postpartum
  Scores from this 34-item scale will be calculated using standard scoring criteria. This scale measures person-centered prenatal care that reflects the experiences of people of color. Scores range from 0 to 100, where higher scores indicate more person-centered prenatal care
Birth satisfaction (BSS-R survey) | After delivery up to 6 weeks postpartum
  Patient satisfaction as measured by the BSS-R with a possible score of 0-40 with 0 equaling the least birth satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Sindhu K Srinivas, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No